CLINICAL TRIAL: NCT00878319
Title: A Randomized Prospective Trial Comparing Operative and Nonoperative Treatment of Humeral Shaft Fractures
Brief Title: Operative and Nonoperative Treatment of Humeral Shaft Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Orthopaedic Trauma Society (Other)
Responsible Party: Principal Investigator, Greg K. Berry, MD, MDCM FRCSC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDR-08-055
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2020-02

CONDITIONS: Humeral Diaphyseal Fracture
Keywords: Humeral; diaphyseal (mid-shaft); fracture; operative; non-operative
MeSH Terms: conditions — Fractures, Bone | interventions — Open Fracture Reduction; Fracture Fixation, Internal; Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical (Active Comparator): Surgical intervention: open reduction and internal fixation (ORIF)
  Interventions: Procedure: Open reduction and internal fixation (ORIF)
- Non-surgical (Active Comparator): Sugartong splint followed by transition to functional co-aptation brace
  Interventions: Other: Non-surgical

INTERVENTIONS:
Procedure: Open reduction and internal fixation (ORIF) — Antero-latero or posterior surgical approach using dynamic compression plate
  Other Names: Plate with locking screws can be used.
  Arms: Surgical
Other: Non-surgical — Sugartong splint followed by transition to functional co-aptation brace
  Arms: Non-surgical

SUMMARY:
The purpose of this research study is to compare two different ways of treating a broken arm (fractured humerus) using either, the nonoperative approach or the operative, open reduction and internal fixation (ORIF). The study will examine which treatment will overall give better results in regards to shoulder and elbow function, residual pain and deformity.

Patients who agree to consent to participation in this study will be randomly selected to receive one of the two treatment methods:

1. Nonoperative: This method requires the application of a plaster sugartong splint for 10 - 14 days followed by a transition to a functional (coaptation) brace to be worn for 4-6 weeks. Patients will be followed by physiotherapy from the baseline visit at 2 weeks.
2. Operative: This treatment option involves an operative procedure for fixation of the broken bone with plates and screws (open reduction internal fixation - ORIF). With this method of treatment, a splint or sling is worn for comfort postoperatively. The patient will be followed by physiotherapy after the post-operative visit at 2 weeks.

Standard follow-up clinic visits at 2 weeks, 6 weeks, 4 months, 6 months and 12 months will be arranged from the date of randomization. The patient will be asked to complete two questionnaires, reporting the level of wellbeing and physical function. These questionnaires will be given to the patient at the time of baseline visit at 2 weeks and again at 6 weeks, 4 months, 6 months and 12 months. They should take approximately 10 - 20 minutes to complete. At each appointment, the patients will be x-rayed until healing has occurred, examined and evaluated (Constant Shoulder Score) by the surgeon and followed by physiotherapy for gentle range of motion (ROM) exercises progressing to strengthening and proprioception of the elbow and shoulder.

DETAILED DESCRIPTION:
Fractures of the humeral diaphysis occur in a bimodal distribution and represent 3-5% of all fractures. Overall the incidence is higher in women and typically presents at a more advanced age in this population, rendering fixation more difficult due to osteoporosis. The majority of fractures of the humeral diaphysis occur in the mid-shaft and proximal third and the majority are simple (or non-comminuted) in pattern.

Presently, the standard treatment of isolated humeral diaphysis fractures is nonoperative care using splints, braces, casts and slings. Most centres in North America and Europe favor functional bracing with a coaptation splint given the positive results reported with this device, despite the prolonged period of pain and discomfort as well as the need for repeated clinic follow-up visits associated with it.

Presently there are no published prospective comparative studies that systematically evaluate patient function following the operative or nonoperative treatment of humeral shaft fractures.

Clinical evaluations following functional bracing using patient-based outcome tools revealed a 20% nonunion rate in patients suffering a simple (non-comminuted) fracture. Invariably, this led to surgical intervention to achieve union. In those whose fracture healed with the splint, only 50% reported a full recovery while none of those requiring surgery for nonunion did so. This low rate of functional recovery may be due in part to the high rate of shoulder stiffness following functional bracing. Significant stiffness in the shoulder following functional bracing has ranged from 14-60% with an average of 40%.

The advantages of open reduction and plate fixation of humeral shaft fractures include a direct approach to the fracture site with direct visualization and protection of the radial nerve (depending on fracture level and approach), the possibility of rigid compressive fixation, and the opportunity for bone grafting and/or radial nerve exploration if needed. Importantly, it permits rapid mobilization of the shoulder and elbow, obviating the need of immobilization, and ensures anatomic or near anatomic alignment. These advantages must be weighed against the small risk of infection (<1-6%) with most occurring after open fractures or severe crush injury, nonunion (4-6%) especially in high energy injuries, and iatrogenic radial nerve injury (1-3%) the vast majority of which are transient.

Operative care: Fixation with regular or broad 3.5mm or 4.5mm dynamic compression plate (DCP) using standard technique will be applied in cases with normal bone density; in the face of osteopenic bone, locked-plate implants will be employed at the discretion of the surgeon. Bone graft will not be used routinely as these are simple fracture patterns. Postoperative splinting (or sling) will be maintained for 10 - 14 days followed by gentle ROM exercises under physiotherapy supervision. Strengthening and proprioception will be begun once fracture healing has occurred, typically at 6-8 weeks.

Conservative care will entail the application of a plaster sugartong splint for 10-14 days followed by transition to a functional (coaptation) brace, to be applied by a qualified orthotist. Gentle ROM exercises of the elbow and shoulder will begin as tolerated under the supervision of a physiotherapist after 2 weeks with strengthening and proprioception added once fracture healing has occurred, typically at 6-8 weeks.

This multicentre prospective randomized trial will involve the Canadian Orthopaedic Trauma Society (COTS), an association of trauma surgeons involved in collaborative outcomes research with a proven track record of research and publication. Patients with a humeral diaphyseal fracture who meet all eligibility criteria and provide consent to participate will be randomly assigned to the operative or splint/brace treatment group. Patients will start physiotherapy at 2 weeks post-randomization (splint/brace group)or 2 weeks post-surgery for gentle ROM exercises. The operative group will progress to strengthening and proprioception at 4-6 weeks. The splint/brace group will only progress at the 6-8 weeks mark once union has occurred. Evaluation at 2 and 6 weeks, 4, 6, and 12 months will include functional, clinical and radiological parameters. Functional evaluation will include the DASH, SMFA questionnaires and the Constant Shoulder Score. Clinical outcome will evaluate range and motion including the shoulder and elbow of both the affected arm and contralateral shoulder and elbow. Standard radiographic parameters will be measured. The primary outcome measure will be functional outcome as measured with the DASH. Appropriate statistical analyses will be performed on the data. Sample size calculation reveals the need for 90 patients per treatment arm. A census of the centers committed to the study predicts a 1-24 month recruitment period. Patient follow-up will end at the 12 month visit.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 y/o with skeletal maturity, and consenting to participate
2. A displaced fracture of the humeral diaphysis amenable to fixation with a plate with no other injuries to the same limb
3. 21 days or less between injury and surgery
4. Medically fit for anaesthesia
5. The mental faculties to participate in post-op evaluation
6. Fracture amenable to both treatment methods

Exclusion Criteria:

1. Open fracture
2. Neurovascular injury requiring repair in the same limb (excluding radial nerve palsy)
3. Active infection in the area of the surgical approach
4. Prior injury, degenerative condition, or congenital condition to the shoulder, arm or elbow
5. Bone disorder which may impair bone healing
6. Polytrauma with other limb fractures
7. Incapable of ensuring follow-up
8. Pathologic fracture
9. Already enrolled in another research clinical trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-08-19 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Validated functional outcome tools to be used: disability shoulder, arm, hand (DASH), short musculoskeletal functional assessment (SMFA) and Constant Shoulder Score. | 2 and 6 weeks, 4, 6 and 12 months

SECONDARY OUTCOMES:
Range of Motion will be measured with a goniometer for both the shoulder/elbow with comparative values taken for a contralateral shoulder/elbow. | 2 and 6 weeks; 4, 6 and 12 months
Radiologic Outcome: Antero-posterior and lateral radiographs | 2 and 6 weeks; 4, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory K. Berry, MDCM FRCSC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre - Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crolla RM, de Vries LS, Clevers GJ. Locked intramedullary nailing of humeral fractures. Injury. 1993 Jul;24(6):403-6. doi: 10.1016/0020-1383(93)90106-g. PMID 8406748
- [Background] Tytherleigh-Strong G, Walls N, McQueen MM. The epidemiology of humeral shaft fractures. J Bone Joint Surg Br. 1998 Mar;80(2):249-53. doi: 10.1302/0301-620x.80b2.8113. PMID 9546454
- [Background] Ekholm R, Adami J, Tidermark J, Hansson K, Tornkvist H, Ponzer S. Fractures of the shaft of the humerus. An epidemiological study of 401 fractures. J Bone Joint Surg Br. 2006 Nov;88(11):1469-73. doi: 10.1302/0301-620X.88B11.17634. PMID 17075092
- [Background] Ekholm R, Tidermark J, Tornkvist H, Adami J, Ponzer S. Outcome after closed functional treatment of humeral shaft fractures. J Orthop Trauma. 2006 Oct;20(9):591-6. doi: 10.1097/01.bot.0000246466.01287.04. PMID 17088659
- [Background] BANDI W. [INDICATION TO AND TECHNIC FOR OSTEOSYNTHESIS IN THE SHOULDER]. Helv Chir Acta. 1964 Jan;31:89-100. No abstract available. German. PMID 14128305
- [Background] Sarmiento A, Waddell JP, Latta LL. Diaphyseal humeral fractures: treatment options. Instr Course Lect. 2002;51:257-69. PMID 12064111
- [Background] Rosenberg N, Soudry M. Shoulder impairment following treatment of diaphysial fractures of humerus by functional brace. Arch Orthop Trauma Surg. 2006 Sep;126(7):437-40. doi: 10.1007/s00402-006-0167-9. Epub 2006 Jun 21. PMID 16810551
- [Background] Koch PP, Gross DF, Gerber C. The results of functional (Sarmiento) bracing of humeral shaft fractures. J Shoulder Elbow Surg. 2002 Mar-Apr;11(2):143-50. doi: 10.1067/mse.2002.121634. PMID 11988725
- [Background] Hunter SG. The closed treatment of fractures of the humeral shaft. Clin Orthop Relat Res. 1982 Apr;(164):192-8. PMID 7067285
- [Background] Ruedi T, Moshfegh A, Pfeiffer KM, Allgower M. Fresh fractures of the shaft of the humerus--conservative or operative treatment? Reconstr Surg Traumatol. 1974;14(0):65-74. No abstract available. PMID 4843035
- [Background] Sarmiento A, Kinman PB, Galvin EG, Schmitt RH, Phillips JG. Functional bracing of fractures of the shaft of the humerus. J Bone Joint Surg Am. 1977 Jul;59(5):596-601. PMID 873955
- [Background] Sarmiento A, Zagorski JB, Zych GA, Latta LL, Capps CA. Functional bracing for the treatment of fractures of the humeral diaphysis. J Bone Joint Surg Am. 2000 Apr;82(4):478-86. doi: 10.2106/00004623-200004000-00003. PMID 10761938
- [Background] Wallny T, Westermann K, Sagebiel C, Reimer M, Wagner UA. Functional treatment of humeral shaft fractures: indications and results. J Orthop Trauma. 1997 May;11(4):283-7. doi: 10.1097/00005131-199705000-00011. PMID 9258827
- [Background] Zagorski JB, Latta LL, Zych GA, Finnieston AR. Diaphyseal fractures of the humerus. Treatment with prefabricated braces. J Bone Joint Surg Am. 1988 Apr;70(4):607-10. PMID 3356728
- [Background] McCormack RG, Brien D, Buckley RE, McKee MD, Powell J, Schemitsch EH. Fixation of fractures of the shaft of the humerus by dynamic compression plate or intramedullary nail. A prospective, randomised trial. J Bone Joint Surg Br. 2000 Apr;82(3):336-9. doi: 10.1302/0301-620x.82b3.9675. PMID 10813165
- [Background] Rockwood CA, Jr, Green DP. Fractures in Adults. Fourth Edition. Philadelphia. Lippincott-Raven, p 1025-53, 1996
- [Background] Chapman JR, Henley MB, Agel J, Benca PJ. Randomized prospective study of humeral shaft fracture fixation: intramedullary nails versus plates. J Orthop Trauma. 2000 Mar-Apr;14(3):162-6. doi: 10.1097/00005131-200003000-00002. PMID 10791665
- [Background] Canadian Orthopaedic Trauma Society. Nonoperative treatment compared with plate fixation of displaced midshaft clavicular fractures. A multicenter, randomized clinical trial. J Bone Joint Surg Am. 2007 Jan;89(1):1-10. doi: 10.2106/JBJS.F.00020. PMID 17200303
- [Background] Buckley R, Tough S, McCormack R, Pate G, Leighton R, Petrie D, Galpin R. Operative compared with nonoperative treatment of displaced intra-articular calcaneal fractures: a prospective, randomized, controlled multicenter trial. J Bone Joint Surg Am. 2002 Oct;84(10):1733-44. doi: 10.2106/00004623-200210000-00001. PMID 12377902
- [Background] Csizy M, Buckley R, Tough S, Leighton R, Smith J, McCormack R, Pate G, Petrie D, Galpin R. Displaced intra-articular calcaneal fractures: variables predicting late subtalar fusion. J Orthop Trauma. 2003 Feb;17(2):106-12. doi: 10.1097/00005131-200302000-00005. PMID 12571499
- [Background] Howard JL, Buckley R, McCormack R, Pate G, Leighton R, Petrie D, Galpin R. Complications following management of displaced intra-articular calcaneal fractures: a prospective randomized trial comparing open reduction internal fixation with nonoperative management. J Orthop Trauma. 2003 Apr;17(4):241-9. doi: 10.1097/00005131-200304000-00001. PMID 12679683
- [Background] Sanders R. Orthopaedic trauma societies and the multicenter trial. J Orthop Trauma. 2006 Jul;20(6):377. doi: 10.1097/00005131-200607000-00001. No abstract available. PMID 16825960
- [Background] Canadian Orthopaedic Trauma Society. Reamed versus unreamed intramedullary nailing of the femur: comparison of the rate of ARDS in multiple injured patients. J Orthop Trauma. 2006 Jul;20(6):384-7. doi: 10.1097/00005131-200607000-00003. PMID 16825962